CLINICAL TRIAL: NCT06804330
Title: Evaluation of Postoperative Pain and Antimicrobial Efficacy of Selenium Versus Calcium Hydroxide As Intracanal Medication in Mandibular First Molars with Necrotic Pulp and Symptomatic Apical Periodontitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Mohamed Wael Mahmoud, Teaching assistant at the department of Endodontics at the faculty of oral and dental medicine, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUE.REC(15)/6-2024
Record Dates: First submitted 2024-08-05; First posted 2025-02-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Necrotic Pulp with Symptomatic Apical Periodontitis; Postoperative Dental Pain; Antimicrobial Effect

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Using Plain Selenium paste as intracanal medication . (Active Comparator)
  Interventions: Procedure: root canal treatment and intracanal medicament
- Using Selenium mixed with calcium hydroxide as intracanal medication . (Active Comparator)
  Interventions: Procedure: root canal treatment and intracanal medicament
- Using Calcium hydroxide as an intracanal medication . (Active Comparator)
  Interventions: Procedure: root canal treatment and intracanal medicament

INTERVENTIONS:
Procedure: root canal treatment and intracanal medicament — Root canal biomechanical preparation followed by intracanal placement of intracanal medicament according to the arm

SUMMARY:
The main rational behind intracanal medicament is to kill the bacteria inside the root canal and to avert reinfection. In absence of nutrients, the bacteria remains after obturation in root canal may not survive. Otherwise they may flourish & If the root canal is not dressed properly with antiseptic medicaments between the visits, the residual bacteria may increase . Thus the use of effective intracanal medication for disinfection of root canal is necessitated . Medicament with long effect and least irritated to periradicular tissue has to be introduced to infiltrate the dentinal tubule eliminating bacteria . As the effect of intracanal medicaments is longer than irrigants, it is generally recommended to fill the root canal between appointments with intracanal medicaments. Calcium hydroxide is the most commonly recommended antimicrobial agent for interappointment medications. It serves as an effective intracanal medicament due to its alkaline pH, which inhibits bacterial growth. However, calcium hydroxide has limitations. .Recently selenium(Se) was introduced as intracanal medication .Se is a mineral essential for the formation of the amino acid selenocysteine, which is directly involved in the maintenance of the immune response. Selenium has been widely used in the medical field in the treatment of cancer, as an activator of bone metabolism, and as a stimulator of the immune system. In this study, it will show that the incorporation of Se, whether as intracanal medication alone or in conjunction with other medications, may potentiate periapical tissue repair after RCS cleaning and shaping procedures.

This study consists of 60 patients divided into 3 group each group having 20 patient.

Intervention 1: intracanal medication using selenium alone .

Intervention 2: intracanal medication using selenium with calcium hydroxide

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients with no systemic disease: (American Society of Anesthesiologists / (ASA Class I or II).

  * Age range is between 20 to 40 years.
  * No sex predilection.
  * Patients having necrotic pulp with symptomatic apical periodontitis in mandibular first molars.(type l distal root canal ) .
  * Sensitive to percussion.
  * Periapical radiographic appearance of teeth showed slight widening in lamina dura.
  * restorable teeth.
  * Positive patient"s acceptance for participating in the study.
  * Patients able to sign informed consent.

Exclusion Criteria:

* Medically compromised patients.

  * Pregnant or lactating females.
  * Psychologically disturbed patients.
  * Patients with a history of allergy to any medication used in the study were excluded.
  * If anti-inflammatory analgesics or antibiotics have been administrated by patient during the past 12 hours preoperatively.
  * Patients with swelling or acute peri-apical abscess or fistulous tract.

Teeth that have:

* Wide or open apex.
* Vital pulp tissues.
* Periodontally affected with grade 2 or 3 mobility.
* Not restorable teeth.
* Abnormal anatomy and calcified canals.
* Previous root canal treatment.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 6 hours up to 96 hours
  Numerical rate scale (NRS) for measuring post-operative pain after 6 hours upto 96 hours 0-10 scale , with zero meaning ''no pain '' and 10 meaning ''the worst pain imaginable ''

SECONDARY OUTCOMES:
Bacterial Load | Before intracanal medication injection and 2 weeks following the procedure and before obturating the root canals
  Serial dilution technique For measuring bacterial load preplacement of the medication and 2 weeks postplacement .

IPD SHARING:
Plan to Share IPD: Undecided